CLINICAL TRIAL: NCT05864469
Title: The Effects of a Psychosocial Dyadic Intervention on the Mutuality, Psychological and Quality of Life Outcomes of Patients With Heart Failure and Their Family Caregivers: A Mixed-methods Study
Brief Title: A Psychosocial Dyadic Programme for Patients With Heart Failure and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Can XIONG, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 23-226
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: dyadic coping; psychosocial intervention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12-week psychosocial dyadic intervention (Experimental): The 12-week psychosocial dyadic intervention will comprise six weekly 60-min telephone-based sessions, followed by two weekly and two bi-weekly telephone follow-ups.
  Interventions: Other: 12-week psychosocial dyadic intervention
- Usual care (No Intervention): Participants in the control group will receive the usual care provided by the clinical team in the hospital

INTERVENTIONS:
Other: 12-week psychosocial dyadic intervention — Comprising six weekly 60-min telephone-based sessions, followed by two weekly and two bi-weekly telephone follow-ups.
  Arms: 12-week psychosocial dyadic intervention

SUMMARY:
The overall aim of the study is to evaluate the effects of a psychosocial dyadic intervention on mutuality, psychological strengths (i.e., resilience and self-compassion), psychological distress (i.e., anxiety and depression), and QoL outcomes of HF patients and caregivers. The HF patient-caregiver dyads will be randomly allocated to the intervention group to receive a 12-week relationship-focused psychosocial dyadic intervention, or to the control group to receive the usual care provided by the clinical team in the hospital.

DETAILED DESCRIPTION:
Heart failure (HF) is the terminal stage of various cardiovascular diseases. HF patient-caregiver dyads, who need to undertake the majority of HF care responsibility in the community, often experience a challenging adaptive process. There is a desperate need to develop and evaluate psychosocial dyadic interventions in HF patients and caregivers, as well as examine the working mechanism of such interventions. This sequential mixed-methods study consists of a single-blinded, two-arm randomized controlled trial (RCT) and a qualitative study. The dyads will be randomly allocated in a 1:1 ratio to the intervention group to receive a 12-week relationship-focused psychosocial dyadic programme, or to the control group to receive the usual care provided by the clinical team in the hospital. Besides, an empowerment-based approach will be employed in this programme to work together with patients and caregivers to set goals and develop an action plan to facilitate goal attainment. For the patients, Mutuality Scale, Connor-Davidson Resilience Scale, Self-Compassion Scale Short Form, Minnesota Living with Heart Failure Questionnaire, and Hospital Anxiety and Depression Scale will be administered at baseline, immediate and 3-month post-intervention. For the caregivers, the Mutuality Scale, Connor-Davidson Resilience Scale, Self-Compassion Scale Short Form, Family Caregiver Quality of Life Scale, and Hospital Anxiety and Depression Scale will be administered at baseline, immediate and 3-month post-intervention. A pilot study will be conducted to determine the feasibility, acceptability and preliminary effect of the intervention first. Afterwards, a full-scale mixed-methods study will be conducted to evaluate the effects of the intervention and the mechanism underlying the intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients and caregivers aged 18 years or older
* patients diagnosed with heart failure
* able to identify one family caregiver who provides unpaid daily caregiving≥3.5hr/ day to participate
* patients and caregivers able to read simplified Chinese and communicate in Mandarin
* have access to a telephone at home.

Exclusion Criteria:

* psychiatric problems requiring active treatment
* other terminal illnesses, such as advanced cancer
* with mechanical circulatory support, on the heart transplant list or with a history of heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Mutuality Scale | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Mutuality Scale (MS, Chinese version) will be used to measure the relationship quality between HF patients and caregivers. The 15-item Mutuality Scale consists of four dimensions: love and affection, shared values, shared enjoyable activities, and reciprocity. The 5-point Likert-type scale from 0 (not at all) to 4 (quite a lot) is used, with higher scores indicating better relationship quality.

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The 10-item Connor-Davidson Resilience Scale (CD-RISC, Chinese version) will be adopted to measure resilience in patients and caregivers. Each item is rated on a 5-point Likert scale from 0 (not true at all) to 4 (true nearly all the time). The scores range from 0 to 40, with higher values implying greater resilience.
Self-Compassion Scale Short Form | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The 12-item Self-Compassion Scale Short Form (SCS-SF, Chinese version) will be used to measure self-compassion in patients and caregivers. Each item is rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always). The score ranges from 12 to 60, with higher scores indicating a higher level of self-compassion.
Minnesota Living with Heart Failure Questionnaire | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Chinese version of the Minnesota Living with Heart Failure Questionnaire (MLHFQ) will be used to measure the disease-specific health-related QoL in HF patients. Patients respond to the 21 items using a 6-point Likert scale (0 = no; 5 = very much). The total score ranges from 0 to 105, with lower scores indicating better health-related QoL.
Family Caregiver Quality of Life Scale | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Chinese version of the Family Caregiver Quality of Life Scale (FAMQoL) will be adopted to measure the QoL in caregivers. The five-point Likert scale with replies ranging from "strongly disagree" to "strongly agree" is used. The total scores range from 16 to 80, and higher scores indicate better QoL.
Hospital Anxiety and Depression Scale | Changes from Baseline at the 3 months (after the intervention) and 6 months (follow-up)
  The Hospital Anxiety and Depression Scale (HADS) was used to evaluate the psychological distress of patients and caregivers. The 4-point Likert scale from 0 (not a problem) to 3 (high level of problems) is applied. The higher scores in the two sub-scales indicate a more intensive anxious and depressed mood.

CONTACTS AND LOCATIONS:
Overall Officials: Can Xiong, PhD student, Principal Investigator — The University of Hong Kong
Locations (1):
- Union hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No